CLINICAL TRIAL: NCT02764255
Title: Does Embryoscope Improve Reproductive Outcome in ICSI Patients
Brief Title: Embryoscope and Reproductive Outcome
Status: Completed | Type: Observational
Sponsor: Ahmed Maged (Other)
Responsible Party: Sponsor-Investigator, Ahmed Maged, Assistant professor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 146
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2016-05

CONDITIONS: Invitro Fertilization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- embryoscope group: cases with embryos continuously monitored by the embryoscope followed by embryo selection based on a multivariable model
- control group: cases with embyos cultured in the standard incubator and evaluated only by morphology

SUMMARY:
cases with embyos cultured in the standard incubator and evaluated only by morphology are compared to cases with embryos continuously monitored by the embryoscope followed by embryo selection based on a multivariable model

DETAILED DESCRIPTION:
cases with embyos cultured in the standard incubator and evaluated only by morphology (control group) are compared to cases with embryos continuously monitored by the embryoscope followed by embryo selection based on a multivariable model(study group)

ELIGIBILITY:
Inclusion Criteria:

* Patient age:25-40 years old
* BMI:18-30
* patients with first or second ICSI trial

Exclusion criteria:

* AMH <1
* severe male factor(total motile sperm <1 million)
* frozen embryo transfer cycles
* patients with endocrinopathies or thrombophilia
* patients on medical treatment which may interfere with results
* hydrosalpinx

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 770 women undergoing ICSI cycles
Sampling Method: Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 14 days after embryo transfer
  transvaginal ultrasound done to assess the gestational sac

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school

IPD SHARING:
Plan to Share IPD: No